CLINICAL TRIAL: NCT01520064
Title: Post Market Registry Study of the AeriSeal System
Status: Terminated | Type: Observational
Sponsor: Aeris Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: 03-C12-001PLV
Record Dates: First submitted 2012-01-25; First posted 2012-01-27 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Pulmonary Emphysema
Keywords: Emphysema; GOLD Stage III; GOLD Stage IV; AeriSeal System; Homogeneous; Heterogeneous; Upper Lobe Predominant; ULP; Chronic Obstructive Pulmonary Disease; COPD; Lung Volume Reduction Surgery; LVRS; Bronchoscopic Lung Volume Reduction; BLVR
MeSH Terms: conditions — Pulmonary Emphysema; Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
* Obtain and analyze medical record data on patients with advanced emphysema who receive treatment with the AeriSeal System to better understand safety and effectiveness in the post-market setting;
* Provide participating physicians access to specified data sets for the purpose of generating scientific manuscripts about the effects of AeriSeal System treatment.

ELIGIBILITY:
Inclusion Criteria:

* Advanced Emphysema
* AeriSeal System treatment

Exclusion Criteria:

* have a primary diagnosis of asthma, chronic bronchitis or bronchiectasis
* have had frequent COPD exacerbations within the past year
* require mechanical ventilatory support
* have a pretreatment DLCO < 20% predicted or > 60% predicted
* have a pretreatment FEV1 < 20% predicted AND homogeneous emphysema
* have giant bullae
* have undergone lung transplantation, lung volume reduction surgery, or lobectomy
* are intolerant of corticosteroids or antibiotics
* are pregnant or breast-feeding

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must have been or will be treated with the AeriSeal System
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Post Market Registry Study of the AeriSeal System | At least 4 years
  -Obtain and analyze medical record data on patients with advanced emphysema who receive treatment with the AeriSeal System to better understand safety and effectiveness in the post-martet setting

CONTACTS AND LOCATIONS:
Overall Officials: Janine McDermott, MS CCRP, Study Director — Aeris Therapeutics
Locations (12):
- Germany (10):
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Klinikum Coburg, Coburg
  - Klinikum Donaustauf, Donaustauf
  - Asklepios Fachkliniken Muenchen-Gauting, Gauting
  - Universitatsklinikum Halle, Halle
  - Asklepios Klinik Hamburg-Harburg, Hamburg
  - Thoraxklinik am Uniklinikum Heidelberg, Heidelberg
  - Sana Kliniken Luebeck, Lübeck
  - Klinikum Nuerberg Nord, Nuremberg
  - Bethanien KH Solingen, Solingen
- Israel (2):
  - Soroka Medical Center, Beer Sheeva
  - Rabin Medical Center, Beilinson Campus, Petach Tikvah